CLINICAL TRIAL: NCT00018057
Title: Study of Neuro-Cognitive Correlates of Pediatric Anxiety Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: University of Minnesota (Other); University of Oregon (Other); University of Maryland (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 010192; 01-M-0192
Record Dates: First submitted 2001-06-29; First posted 2001-07-02 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-09

CONDITIONS: Anxiety Disorders; Major Depressive Disorder
Keywords: fMRI; Emotion; Normal Volunteers; Magnetic Resonance Imaging; CBT
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Subjects in both treatment arms receive cognitive behavioral therapy (CBT) for a 12-week period. In the final eight weeks of the trial, the subjects complete either the active-intervention arm or the control invention arm. In these arms, either the active or control treatment is administered immediately before a CBT session.
  Interventions: Behavioral: Attention Bias Modification Training; Drug: Fluoxetine
- Control (Placebo Comparator): Subjects in both treatment arms receive cognitive behavioral therapy (CBT) for a 12-week period. In the final eight weeks of the trial, the subjects complete either the active-intervention arm or the control invention arm. In these arms, either the active or control treatment is administered immediately before a CBT session.
  Interventions: Behavioral: Attention Bias Modification Training

INTERVENTIONS:
Behavioral: Attention Bias Modification Training — The intervention is computer-based. The active and control treatments have two components. In one component of the active intervention, subjects are asked to indicate the identity of a letter that appears behind a neutral face, opposite from an angry face. In another component of the active intervention, subjects are asked to identify numbers that are hidden within a puzzle, in locations distal from angry faces. In both components of the active intervention, subjects implicitly learn to shift their attention away from angry faces. This is because the faces are systematically arranged to be far removed from letters and numbers that need to be identified. The control arm of the intervention involves similar components. However, unlike in the intervention arm, angry faces appear in various locations near letters and numbers. Therefore, attention is not shaped in the control arm. This intervention requires five minutes per session and is administered before weekly psychotherapy sessions.
Drug: Fluoxetine — Randomized assignment.
  Arms: Active

SUMMARY:
Study Description:

This study examines relations between neurocognitive and clinical features of pediatric anxiety disorders. The study uses neuro-cognitive tasks, functional magnetic resonance imaging (fMRI), as well as magneto- and electro-encephalography (M/EEG). Patients will be studied over one year, before and after receiving either one of two standard-of-care treatments: cognitive behavioral therapy (CBT) or fluoxetine, a serotonin reuptake inhibitor (SSRI). Healthy comparisons will be studied at comparable time points.

Primary Objectives:

To compare healthy youth and symptomatic, medication-free pediatric patients studied prior to receipt of treatment. The study seeks to detect relations between clinical features of anxiety disorders at baseline and a wide range of neurocognitive features associated with attention, memory, and response to motivational stimuli.

Secondary Objectives:

1. To document relations between baseline neurocognitive features and response to Cognitive Behavioral Therapy (CBT) or fluoxetine, as defined by the Pediatric Anxiety Rating Scale (PARS) and Clinical Global Improvement (CGI) Scale.
2. To document relations between post-treatment changes in neurocognitive features and anxiety symptoms on the PARS following treatment with Cognitive Behavioral Therapy (CBT) or fluoxetine.
3. To document relations among broad arrays of clinical, cognitive, and neural measures

Primary Endpoints:

Indices of percent-signal change in hypothesized brain regions, comprising amygdala, striatum, and prefrontal cortex (PFC) for each fMRI and MEG paradigm.

Secondary Endpoints:

1. Treatment-response as defined by a continuous measure, the Pediatric Anxiety Rating Scale score (PARS), and a categorial measure, the Clinical Global Improvement (CGI) score.
2. Levels of symptoms and behaviors evoked by tasks that engage attention, memory, and elicit responses to motivational stimuli.

   ...

DETAILED DESCRIPTION:
Study Description:

This study examines relations between neurocognitive and clinical features of pediatric anxiety disorders. The study uses neurocognitive tasks, functional magnetic resonance imaging (fMRI), as well as magneto- and electro-encephalography (M/EEG). Patients will be studied over one year, before and after receiving either one of two standard-of-care treatments: cognitive behavioral therapy (CBT) or fluoxetine, a serotonin reuptake inhibitor (SSRI). Healthy comparisons will be studied at comparable time points.

Primary Objectives:

-To compare healthy youth and symptomatic, medication-free pediatric patients studied prior to receipt of treatment. The study seeks to detect relations between clinical features of anxiety disorders at baseline and a wide range of neurocognitive features associated with attention, memory, and response to motivational stimuli.

Secondary Objectives:

* To document relations between baseline neurocognitive features and response to Cognitive Behavioral Therapy (CBT) or fluoxetine, as defined by the Pediatric Anxiety Rating Scale (PARS) and Clinical Global Improvement (CGI) Scale.
* To document relations between post-treatment changes in neurocognitive features and anxiety symptoms on the PARS following treatment with Cognitive Behavioral Therapy (CBT) or fluoxetine.
* To document relations among broad arrays of clinical, cognitive, and neural measures

Primary Endpoints:

-Indices of percent-signal change in hypothesized brain regions, comprising amygdala, striatum, and prefrontal cortex (PFC) for each fMRI and MEG paradigm.

Secondary Endpoints:

* Treatment-response as defined by a continuous measure, the Pediatric Anxiety Rating Scale score (PARS), and a categorial measure, the Clinical Global Improvement (CGI) score.
* Levels of symptoms and behaviors evoked by tasks that engage attention, memory, and elicit responses to motivational stimuli.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALL JUVENILE SUBJECTS

* Age: 8-17 (subjects who consent as 17-year-olds but turn 18 during the course of the study will be eligible to complete all procedures completed by other subjects who consent as 17-year-olds but do not turn 18).
* Consent: can give consent/assent (Parents will provide consent; minors will provide assent)
* IQ: all subjects will have IQ>70 (Assessment relies on either a WASI or assessment by trained clinical staff during the subject s screening visit. Completion of required activities during the screening visit requires an IQ above 70.)
* Language: all subjects will speak English (Tasks in this protocol have not been validated in languages other than English)

ALL ADULT SUBJECTS

* Age: 18-65
* Consent: can give consent
* IQ: all subjects will have IQ>70 (Assessment relies on either a WASI or assessment by trained clinical staff during the subject s screening visit. Completion of required activities during the screening visit requires an IQ above 70.)
* Language: all subjects will speak English (Tasks in this protocol have not been validated in languages other than English)

ALL SUBJECTS WITH AN ANXIETY DISORDER

* Diagnosis: Current Diagnosis of Social Phobia, Separation Anxiety, Generalized Anxiety Disorder, or Panic Disorder (Based on K-SADS (juveniles) or SCID (adults))
* Symptom Severity: Clinically significant, ongoing anxiety symptoms (This will be documented by clinician review with patients and their families during at least two visits with families.)
* Clinical Impairment: Clinically significant, ongoing distress or impairment from anxiety (This will be documented by clinician review with patients and their families during at least two visits with families.)

ALL PREVIOUSLY ENROLLED ADOLESCENT PATIENTS, CHILD AND ADULT HEALTHY VOLUNTEERS, AND ALL HEALTHY VOLUNTEERS TURNED PATIENTS

* Diagnosis: Current Diagnosis of Social Phobia, Separation Anxiety, Generalized Anxiety Disorder, or Panic Disorder; No current diagnosis (Based on K-SADS (juveniles) or SCID (adults))
* Clinical Impairment (as applicable): Clinically significant, ongoing symptoms (This will be documented by clinician review with patients and their families during at least two visits with families.)
* Symptom Severity (as applicable): Clinically significant, ongoing symptoms (This will be documented by clinician review with patients and their families during at least two visits with families.)

EXCLUSION CRITERIA:

ALL SUBJECTS

* Any serious medical condition or condition that interferes with fMRI or M/EEG scanning, and for patients electing medication, any condition that increases risk of SSRI treatment. (All patients will complete a medical history. Healthy volunteer participants will be medication- free and have no current serious medical conditions, based on a review of their medical history. Subjects only will be excluded from the MRI portions of the study based on this exclusion criterion.)
* Pregnancy (Subjects only will be excluded from the MRI portions of the study based on this exclusion criterion.)
* Current use of any psychoactive substance; current suicidal ideation; current diagnosis of attention deficit hyperactivity disorder (ADHD) of sufficient severity to require pharmacotherapy. (These factors could complicate treatment with an SSRI. No subject on medication will be accepted into the trial. Subjects will not be taken off of medications to enter the trial.)
* Current diagnoses Tourette's Disorder, major depressive disorder (MDD); obsessive compulsive disorder (OCD), post-traumatic distress disorder, conduct disorder. (These factors may be affected by SSRI treatment, influencing ability to detect effects on anxiety/symptoms of depression. Of note, subjects who present with a diagnosis of MDD or OCD will not be eligible for inclusion at the outset of the study. However, youth with anxiety disorders frequently develop OCD and MDD when followed over time. Subjects will be allowed to remain in the study if they develop these diagnoses after enrollment.)
* Past or current history of mania, psychosis, or severe pervasive developmental disorder. (These factors may be affected by SSRI treatment, influencing ability to detect effects on anxiety/symptoms of depression. Of note, subjects who present with a diagnosis of MDD or OCD will not be eligible for inclusion at the outset of the study. However, youth with anxiety disorders frequently develop OCD and MDD when followed over time. Subjects will be allowed to remain in the study if they develop these diagnoses after enrollment.)
* Recent use of an SSRI with failure to respond or tolerate SSRI treatment at an adequate dose and duration. (This is designed to exclude subjects who have failed a trial of an SSRI for their current problem with anxiety. For previously enrolled participants, including patients and healthy volunteers, current use of an SSRI does not exclude participation from follow-up research tasks.)
* History of any (excepting nicotine-related and cannabis-related) DSM5-defined moderate to severe substance use disorder (or DSM-IV-defined substance dependence).

HEALTHY ADULT SUBJECTS

-Any current psychiatric diagnosis (Assessment relies on SCID)

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2530 (Estimated)
Dates: Start 2001-10-02 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale (PARS) | Weekly
  Clinician-rated report
Clinical Global Improvement (CGI) Scale | Weekly
  Clinician-rated report

SECONDARY OUTCOMES:
Another secondary objective is to document relations between post-treatment changes in neurocognitive features and anxiety symptoms on the PARS following treatment with Cognitive Behavioral Therapy (CBT) or fluoxetine. | Changes in symptoms on PARS and changes after 8-12 weeks of treatment in patients
  Prior research in adults finds changes in symptoms to relate to changes in brain function. If confirmed in youth, this would provide insights on mechanisms of therapeutic change and targets for novel therapies

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Byrne ME, Bernstein RA, Pine DS, Kircanski K. Ecological Momentary Assessment of Youth Anxiety: Evaluation of Psychometrics for Use in Clinical Trials. J Child Adolesc Psychopharmacol. 2023 Dec;33(10):409-417. doi: 10.1089/cap.2023.0025. Epub 2023 Dec 5. PMID 38052059
- [Derived] Tseng WL, Naim R, Chue A, Shaughnessy S, Meigs J, Pine DS, Leibenluft E, Kircanski K, Brotman MA. Network analysis of ecological momentary assessment identifies frustration as a central node in irritability. J Child Psychol Psychiatry. 2023 Aug;64(8):1212-1221. doi: 10.1111/jcpp.13794. Epub 2023 Mar 28. PMID 36977629
- [Derived] Linke JO, Haller SP, Xu EP, Nguyen LT, Chue AE, Botz-Zapp C, Revzina O, Perlstein S, Ross AJ, Tseng WL, Shaw P, Brotman MA, Pine DS, Gotts SJ, Leibenluft E, Kircanski K. Persistent Frustration-Induced Reconfigurations of Brain Networks Predict Individual Differences in Irritability. J Am Acad Child Adolesc Psychiatry. 2023 Jun;62(6):684-695. doi: 10.1016/j.jaac.2022.11.009. Epub 2022 Dec 21. PMID 36563874
- [Derived] Newsome P, Ruiz SG, Gold AL, Pine DS, Abend R. Fear-potentiated startle reveals diminished threat extinction in pathological anxiety. Int J Psychophysiol. 2023 Jan;183:81-91. doi: 10.1016/j.ijpsycho.2022.11.011. Epub 2022 Nov 25. PMID 36442665
- [Derived] Naim R, Shaughnessy S, Smith A, Karalunas SL, Kircanski K, Brotman MA. Real-time assessment of positive and negative affective fluctuations and mood lability in a transdiagnostic sample of youth. Depress Anxiety. 2022 Dec;39(12):870-880. doi: 10.1002/da.23293. Epub 2022 Nov 3. PMID 36325887
- [Derived] Haller SP, Archer C, Jeong A, Jaffe A, Jones EL, Harrewijn A, Naim R, Linke JO, Stoddard J, Brotman MA. Changes in Internalizing Symptoms During the COVID-19 Pandemic in a Transdiagnostic Sample of Youth: Exploring Mediators and Predictors. Child Psychiatry Hum Dev. 2024 Feb;55(1):206-218. doi: 10.1007/s10578-022-01382-z. Epub 2022 Jul 6. PMID 35794298
- [Derived] Scheinost D, Dadashkarimi J, Finn ES, Wambach CG, MacGillivray C, Roule AL, Niendam TA, Pine DS, Brotman MA, Leibenluft E, Tseng WL. Functional connectivity during frustration: a preliminary study of predictive modeling of irritability in youth. Neuropsychopharmacology. 2021 Jun;46(7):1300-1306. doi: 10.1038/s41386-020-00954-8. Epub 2021 Jan 21. PMID 33479511
- [Derived] Cardinale EM, Freitag GF, Brotman MA, Pine DS, Leibenluft E, Kircanski K. Phasic Versus Tonic Irritability: Differential Associations With Attention-Deficit/Hyperactivity Disorder Symptoms. J Am Acad Child Adolesc Psychiatry. 2021 Dec;60(12):1513-1523. doi: 10.1016/j.jaac.2020.11.022. Epub 2021 Jan 10. PMID 33440203
- [Derived] Linke JO, Abend R, Kircanski K, Clayton M, Stavish C, Benson BE, Brotman MA, Renaud O, Smith SM, Nichols TE, Leibenluft E, Winkler AM, Pine DS. Shared and Anxiety-Specific Pediatric Psychopathology Dimensions Manifest Distributed Neural Correlates. Biol Psychiatry. 2021 Mar 15;89(6):579-587. doi: 10.1016/j.biopsych.2020.10.018. Epub 2020 Nov 9. PMID 33386133
- [Derived] Smith AR, Haller SP, Haas SA, Pagliaccio D, Behrens B, Swetlitz C, Bezek JL, Brotman MA, Leibenluft E, Fox NA, Pine DS. Emotional distractors and attentional control in anxious youth: eye tracking and fMRI data. Cogn Emot. 2021 Feb;35(1):110-128. doi: 10.1080/02699931.2020.1816911. Epub 2020 Sep 21. PMID 32954946
- [Derived] Filippi CA, Sachs JF, Phillips D, Winkler A, Gold AL, Leibenluft E, Pine DS, Fox NA. Infant behavioral reactivity predicts change in amygdala volume 12 years later. Dev Cogn Neurosci. 2020 Apr;42:100776. doi: 10.1016/j.dcn.2020.100776. Epub 2020 Mar 21. PMID 32452462
- [Derived] Haller SP, Kircanski K, Stringaris A, Clayton M, Bui H, Agorsor C, Cardenas SI, Towbin KE, Pine DS, Leibenluft E, Brotman MA. The Clinician Affective Reactivity Index: Validity and Reliability of a Clinician-Rated Assessment of Irritability. Behav Ther. 2020 Mar;51(2):283-293. doi: 10.1016/j.beth.2019.10.005. Epub 2019 Nov 27. PMID 32138938
- [Derived] Smith AR, Nelson EE, Kircanski K, Rappaport BI, Do QB, Leibenluft E, Pine DS, Jarcho JM. Social anxiety and age are associated with neural response to social evaluation during adolescence. Dev Cogn Neurosci. 2020 Apr;42:100768. doi: 10.1016/j.dcn.2020.100768. Epub 2020 Feb 10. PMID 32077442
- [Derived] Abend R, Gold AL, Britton JC, Michalska KJ, Shechner T, Sachs JF, Winkler AM, Leibenluft E, Averbeck BB, Pine DS. Anticipatory Threat Responding: Associations With Anxiety, Development, and Brain Structure. Biol Psychiatry. 2020 May 15;87(10):916-925. doi: 10.1016/j.biopsych.2019.11.006. Epub 2019 Nov 15. PMID 31955915
- [Derived] Filippi CA, Subar AR, Sachs JF, Kircanski K, Buzzell G, Pagliaccio D, Abend R, Fox NA, Leibenluft E, Pine DS. Developmental pathways to social anxiety and irritability: The role of the ERN. Dev Psychopathol. 2020 Aug;32(3):897-907. doi: 10.1017/S0954579419001329. PMID 31656217
- [Derived] Abend R, Rosenfelder A, Shamai D, Pine DS, Tavor I, Assaf Y, Bar-Haim Y. Brain structure changes induced by attention bias modification training. Biol Psychol. 2019 Sep;146:107736. doi: 10.1016/j.biopsycho.2019.107736. Epub 2019 Jul 25. PMID 31352029
- [Derived] Cardinale EM, Kircanski K, Brooks J, Gold AL, Towbin KE, Pine DS, Leibenluft E, Brotman MA. Parsing neurodevelopmental features of irritability and anxiety: Replication and validation of a latent variable approach. Dev Psychopathol. 2019 Aug;31(3):917-929. doi: 10.1017/S095457941900035X. Epub 2019 May 8. PMID 31064595
- [Derived] Cardinale EM, Subar AR, Brotman MA, Leibenluft E, Kircanski K, Pine DS. Inhibitory control and emotion dysregulation: A framework for research on anxiety. Dev Psychopathol. 2019 Aug;31(3):859-869. doi: 10.1017/S0954579419000300. Epub 2019 Apr 10. PMID 30968800
- [Derived] Abend R, Swetlitz C, White LK, Shechner T, Bar-Haim Y, Filippi C, Kircanski K, Haller SP, Benson BE, Chen G, Leibenluft E, Fox NA, Pine DS. Levels of early-childhood behavioral inhibition predict distinct neurodevelopmental pathways to pediatric anxiety. Psychol Med. 2020 Jan;50(1):96-106. doi: 10.1017/S0033291718003999. Epub 2019 Jan 8. PMID 30616705
- [Derived] Tseng WL, Deveney CM, Stoddard J, Kircanski K, Frackman AE, Yi JY, Hsu D, Moroney E, Machlin L, Donahue L, Roule A, Perhamus G, Reynolds RC, Roberson-Nay R, Hettema JM, Towbin KE, Stringaris A, Pine DS, Brotman MA, Leibenluft E. Brain Mechanisms of Attention Orienting Following Frustration: Associations With Irritability and Age in Youths. Am J Psychiatry. 2019 Jan 1;176(1):67-76. doi: 10.1176/appi.ajp.2018.18040491. Epub 2018 Oct 19. PMID 30336704
- [Derived] Smith AR, Nelson EE, Rappaport BI, Pine DS, Leibenluft E, Jarcho JM. I Like Them...Will They Like Me? Evidence for the Role of the Ventrolateral Prefrontal Cortex During Mismatched Social Appraisals in Anxious Youth. J Child Adolesc Psychopharmacol. 2018 Nov;28(9):646-654. doi: 10.1089/cap.2017.0142. Epub 2018 May 24. PMID 29792726
- [Derived] Kircanski K, White LK, Tseng WL, Wiggins JL, Frank HR, Sequeira S, Zhang S, Abend R, Towbin KE, Stringaris A, Pine DS, Leibenluft E, Brotman MA. A Latent Variable Approach to Differentiating Neural Mechanisms of Irritability and Anxiety in Youth. JAMA Psychiatry. 2018 Jun 1;75(6):631-639. doi: 10.1001/jamapsychiatry.2018.0468. PMID 29625429
- [Derived] White LK, Sequeira S, Britton JC, Brotman MA, Gold AL, Berman E, Towbin K, Abend R, Fox NA, Bar-Haim Y, Leibenluft E, Pine DS. Complementary Features of Attention Bias Modification Therapy and Cognitive-Behavioral Therapy in Pediatric Anxiety Disorders. Am J Psychiatry. 2017 Aug 1;174(8):775-784. doi: 10.1176/appi.ajp.2017.16070847. Epub 2017 Apr 14. PMID 28407726
- [Derived] Gold AL, Jarcho JM, Rosen DK, Pine DS, Ernst M. Emotional and Nonemotional Conflict Processing in Pediatric and Adult Anxiety Disorders. J Child Adolesc Psychopharmacol. 2015 Dec;25(10):754-63. doi: 10.1089/cap.2015.0066. Epub 2015 Nov 6. PMID 26544668
- [Derived] Britton JC, Suway JG, Clementi MA, Fox NA, Pine DS, Bar-Haim Y. Neural changes with attention bias modification for anxiety: a randomized trial. Soc Cogn Affect Neurosci. 2015 Jul;10(7):913-20. doi: 10.1093/scan/nsu141. Epub 2014 Oct 24. PMID 25344944
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-M-0192.html